CLINICAL TRIAL: NCT00317018
Title: Implementing Telemedicine-Based Collaborative Care for MDD in Contract CBOCs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn prior to enrollment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMV 04-360
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Depression
Keywords: depression; quality improvement; implementation; translation; evidence-based practice; collaborative care; adoption; sustainability; cost-effectiveness; rural
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other): Implementation Group
  Interventions: Behavioral: Evidence-Based Quality Improvement
- Arm 2 (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Evidence-Based Quality Improvement — The implementation intervention is known as Evidence-Based Quality Improvement (EBQI). EBQI is an adaptation of the Plan-Do-Study-Act cycles of Continuous Quality Improvement that emphasizes empirical evidence and the involvement of clinical and implementation experts (i.e., researchers). In the EBQI implementation intervention, both researchers (clinical and implementation experts) and local staff participate fully in the quality improvement process, with the researchers facilitating rather than dictating implementation efforts. Using EBQI methods, researchers and local staff adapt evidence-based practices for local resources, needs and preferences while maintaining fidelity to the evidence-base. PDSA cycles are used to continuously revise the adapted evidence-based practice based on feedback during pilot tests.
  Arms: Arm 1

SUMMARY:
Small contract VA Community Based Outpatient Clinics present unique challenges to implementation of collaborative care because of their distinct organizational characteristics and lack of on-site psychiatrists. A recent effectiveness study, successfully used telemedicine technologies to adapt the collaborative care model for small rural VA Community Based Outpatient Clinics. The purpose of the proposed study is to implement this telemedicine-based collaborative care model in small Contract VA Community Based Outpatient Clinics and determine its sustainability and cost-effectiveness.

DETAILED DESCRIPTION:
Rationale and Objectives: Implementation of collaborative care for depression is the highest priority for Mental Health QUERI, and preparing for national rollout of collaborative care is a key component of the VHA's Mental Health Strategic Plan. In addition, both the Mental Health Task Force Report and the CARES Commission Report have prioritized the provision of mental health services in all CBOCs. Secretary Principi has repeatedly emphasized the importance of this recommendation. However, small Contract CBOCs present unique challenges to implementation of collaborative care because of their distinct organizational characteristics, long distances to parent VAMCs, and lack of onsite psychiatrists. The Telemedicine Enhanced Antidepressant Management (TEAM) study, successfully used telemedicine technologies to adapt the collaborative care model for small CBOCs lacking onsite psychiatrists. The purpose of the proposed RIPPLE study is to implement and evaluate this telemedicine-based collaborative care model in small Contract CBOCs. The goals and aims of the RIPPLE study are:

Goal 1 To adapt and apply implementation strategies developed for TIDES/RETIDES in order to deliver telemedicine-based collaborative care services in small contract CBOCs.

Goal 2: To evaluate the implementation of this evidence-based best-practice with respect to its clinical impact on the population of patients with MDD and the system of care. The corresponding specific aims are:

Specific Aim 1: Document and evaluate the process of implementing, refining, and sustaining telemedicine-based collaborative care at contract CBOCs.

Specific Aim 2: Estimate the clinical impact of telemedicine-based collaborative care at implementation sites relative to usual care at control sites.

Specific Aim 3: Estimate the system-level cost-effectiveness of telemedicine-based collaborative care at contract CBOCs.

Research Design and Study Setting: The study will be conducted in 26 contract CBOCs in VISN 16 and VISN 22. The analyses will be based on a pre-post quasi-experimental study design with a non-equivalent control group. The telemedicine-based collaborative care program will be implemented at 11 contract CBOCs without onsite psychiatrists and cost/outcomes will be compared to those at 15 similar control sites.

Data Collection and Analysis: Data will be collected from survey, key informant interviews, VISTA, and the Austin Automation Center. Descriptive statistics will be used to describe the degree of adoption (i.e., reach, effectiveness, adoption, implementation, and maintenance). The clinical impact on the patient population will be estimated using random effects models with individual patients as the unit of analysis. The impact on the system will be estimated using a Systems Cost Effectiveness Analysis.

Significance: Evaluating strategies for implementing telemedicine-based collaborative care in contract CBOCs should be a high priority for VA for several reasons. First, VA's Mental Health Strategic Plan includes plans for the rollout of collaborative care throughout the entire VA health care system. Second, the importance of providing mental health services in all CBOCs is highlighted by the recent introduction of a performance measure targeting mental health in CBOCs. Third, there are 183 contract CBOCs in the VA health care system, most of which have no on-site psychiatrists and are located in rural areas far from parent VAMCs. Fourth, the TEAM collaborative care model has been demonstrated to significantly and substantially improve depression outcomes in these small rural CBOCs. While the implementation of collaborative care in large VA-staffed clinics is an immensely challenging task, implementing collaborative care in small contract clinics is even more challenging. To prepare for national rollout, it is imperative that implementation strategies be developed and evaluated for these difficult settings in order to avoid the creation of a two-tiered system of care. National rollout strategies must target contract CBOCs to ensure access to collaborative care for all veterans and to prevent future health disparities. In addition, the results of the RIPPLE study will provide a template for the development of best-practice implementation strategies targeting other high priority QUERI disorders in contract CBOCs.

ELIGIBILITY:
Inclusion Criteria:

* veteran
* depression
* patient at Little Rock VAMC, Loma Linda VAMC, or Greater Los Angeles VAMC

Exclusion Criteria:

* veteran
* depression
* patient at Little Rock VAMC, Loma Linda VAMC, or Greater Los Angeles VAMC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reach, Effectiveness, Adoption, Implementation, and Maintenance, percent screening positive for depression, specialty mental health visits, antidepressant medication possession ratio, VA depression performance measure | 12 months

SECONDARY OUTCOMES:
cost-effectiveness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fortney, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System (North Little Rock)
Locations (2):
- United States (2):
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California

REFERENCES:
- [Result] Fortney JC, Pyne JM, Smith JL, Curran GM, Otero JM, Enderle MA, McDougall S. Steps for implementing collaborative care programs for depression. Popul Health Manag. 2009 Apr;12(2):69-79. doi: 10.1089/pop.2008.0023. PMID 19320606
- [Result] Fortney JC, Enderle MA, Clothier JL, Otero JM, Williams JS, Pyne JM. Population level effectiveness of implementing collaborative care management for depression. Gen Hosp Psychiatry. 2013 Sep-Oct;35(5):455-60. doi: 10.1016/j.genhosppsych.2013.04.010. Epub 2013 May 30. PMID 23725825
- [Result] Fortney JC, Pyne JM, Steven CA, Williams JS, Hedrick RG, Lunsford AK, Raney WN, Ackerman BA, Ducker LO, Bonner LM, Smith JL. A Web-based clinical decision support system for depression care management. Am J Manag Care. 2010 Nov;16(11):849-54. PMID 21348556
- [Result] Fortney J, Enderle M, McDougall S, Clothier J, Otero J, Altman L, Curran G. Implementation outcomes of evidence-based quality improvement for depression in VA community based outpatient clinics. Implement Sci. 2012 Apr 11;7:30. doi: 10.1186/1748-5908-7-30. PMID 22494428